CLINICAL TRIAL: NCT03855072
Title: Patient Satisfaction Following Vertical Ramus Osteotomy After Mandibular Setback Fixed With Patients Specific Osteosynthesis and Immediate Mobilization Versus Vertical Ramus Osteotomy Fixed With MMFin Patients With Mandibular Prognanthism
Brief Title: Patient Satisfaction Vertical Ramus Osteotomy Patient Specificosteosynthesis Fixation Versus MMFmandibular Prognanthism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Sayed Abbass Ali, associate lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Goal NO 5 , OMFS IV A3
Record Dates: First submitted 2019-02-21; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Mandibular Prognathism
Keywords: Mandibular Prognanthism,customized plate
MeSH Terms: conditions — Malocclusion, Angle Class III | interventions — Jaw Fixation Techniques

STUDY DESIGN:
Intervention Model Description: * A Randomized Controlled Trial
  * A Trial will be carried out in Hospital of Oral and Maxillofacial surgery departement- faculty of Dentistry , Cairo University
  * Equal randomization : participant with equal probabilities for intervention
  * Parallel group study : Each group of patients recieves a single treatment simultaneously
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Customized plate fixation (Experimental): Customized Plate fixation of Vertical Ramus Osteotomy after Mandibular Setback
  - intervention:
  * All cases will undergo one surgery under general anesthesia.
  * Incision was made medial to external oblique ridge from the asendindg ramus to second molar region
  * The intraoral vertical osteotomy is accomplished by using an oscillating saw to make the cut from the sigmoid notch through the inferior border of the mandible.
  * 3D virtual planning and 3D mandible model represented fom CBCT in MIMICS
  * The customized fixation plate is positioned to fix the proximal and distal segment together
  Interventions: Procedure: customized fixation plate
- maxillomandibular fixation (Active Comparator): Mandibular Setback by Vertical Ramus Ostotmy fixed with Maxillomandibular fixation
  - intervention:
  * All cases will undergo one surgery under general anesthesia
  * incision was made medial to external oblique ridge from the asendindg ramus to second molar region .
  * The intraoral vertical osteotomy is accomplished by using an oscillating saw to make the cut from the sigmoid notch through the inferior border of the mandible.
  * Patient is placed in maxillomandibular fixation (MMF) using a prefabricated occlusal splint
  Interventions: Procedure: maxillomandibular fixation

INTERVENTIONS:
Procedure: customized fixation plate — * All cases will undergo one surgery under general anesthesia.
  * Incision was made medial to external oblique ridge from the asendindg ramus to second molar region
  * Amucoperiosteal flap was reflected to expose the lateral mandibular ramus to the posterior border and the sigmoid notch
  * The intraoral vertical osteotomy is accomplished by using an oscillating saw to make the cut from the sigmoid notch through the inferior border of the mandible.
  * 3D virtual planning and 3D mandible model represented fom CBCT in MIMICS
  * The customized fixation plate is positioned to fix the proximal and distal segment together after setback
  Other Names: patient specific osteosynthesis
  Arms: Customized plate fixation
Procedure: maxillomandibular fixation — * All cases will undergo one surgery under general anesthesia.
  * incision was made medial to external oblique ridge from the asendindg ramus to second molar region .
  * The intraoral vertical osteotomy is accomplished by using an oscillating saw to make the cut from the sigmoid notch through the inferior border of the mandible.
  * Patient is placed in maxillomandibular fixation (MMF) using a prefabricated occlusal splint to assure accuracy of the mandibular position.
  Other Names: intermaxillary fixation
  Arms: maxillomandibular fixation

SUMMARY:
Two groups with mandibular prognanthism indicated for mandibular setback by intraoral vertical ramus osteotomy . first group will fixed with maxillomandibular fixation and the second group will fixed by customized plate

DETAILED DESCRIPTION:
Two groups with mandibular prognanthism indicated for mandibular setback by intraoral vertical ramus osteotomy . first group will fixed with maxillomandibular fixation and the second group will fixed by customized plate

Interventions:

General operative procedures

Eligible patients will be randomized in equal proportions between the study group (customized plate fixation of VRO) and the control group (maxillomandibular fixation of VRO).

Patients of Both groups will be subjected to:

1. Case history including personal data, medical, surgical history and family history
2. Clinical examination .
3. Radiographic examination in the form of cephalometric radiogragh .
4. Preoperative laboratory tests (complete blood cell count, Hemoglobin count, coagulation profile, liver function, kidney function and blood glucose level).
5. Preoperative anesthesia assessment for fitness for general anesthesia.

vertical ramus osteotmy fixed with customized plate

* All cases will undergo one surgery under general anesthesia.
* Incision was made medial to external oblique ridge from the asendindg ramus to second molar region
* Amucoperiosteal flap was reflected to expose the lateral mandibular ramus to the posterior border and the sigmoid notch
* The intraoral vertical osteotomy is accomplished by using an oscillating saw to make the cut from the sigmoid notch through the inferior border of the mandible. The osteotomy is placed 5 mm anterior to the posterior border of the mandible to avoid injury to the inferior alveolar neurovascular bundle
* 3D virtual planning and 3D mandible model represented fom CBCT in MIMICS
* The setback will be simulated according to pre-planned measure
* The customized bone plate is positioned to fix the proximal and distal segment together

vertical ramus osteotomy fixed with MMF.

* All cases will undergo one surgery under general anesthesia.
* incision was made medial to external oblique ridge from the asendindg ramus to second molar region .
* Amucoperiosteal flap was reflected to expose the lateral mandibular ramus to the posterior border and the sigmoid notch
* The intraoral vertical osteotomy is accomplished by using an oscillating saw to make the cut from the sigmoid notch through the inferior border of the mandible. The osteotomy is placed 5 mm anterior to the posterior border of the mandible to avoid injury to inferior alveolar neurovascular bundle.
* Patient is placed in maxillomandibular fixation (MMF) using a prefabricated occlusal splint to assure accuracy of the mandibular position.

follow up clinical and radiographic evaluation will be performed at the first week postoperative then the patients will recalled for radiograghic evaluation at 2weeks and 2 months .finall follow up visit will be at 6 months postoperative

ELIGIBILITY:
Inclusion Criteria:

All subjects were required:

* Patients with mandibular prognanthism indicated for mandibular setback.
* All ages >18 years
* Patients should be free from any systemic disease that may affect normal healing of bone, and predictable outcome.
* Patients with good general condition allowing surgical procedure under general anesthesia.
* Patients with physical and psychological tolerance

Exclusion Criteria:

* History of mandibular trauma
* Previous orthognathic surgery
* Degenerative disease of temporomandibular joint
* Craniofacial syndrome such as cleft lip or palate
* Follow up period will be less than 6 months

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | immediately postoperative
  Patient were asked to fill out a questionnaire in order to investigate their satisfaction degree after surgery ,according to an adapted (10 cm) visual analogue scale (VAS) from 0 to +10 0 is the least satisfied 10 is the most satisfied

SECONDARY OUTCOMES:
stability of Mandible | pre- operative , 2 weeks postoperative , 2 months postoperative , 6 months postoperative
  assessed by determining the differences between measurements of three mandibular reference points (B-point, menton, and pogonion) in relation to SNy ,SNx axis obtained at six different time points